CLINICAL TRIAL: NCT05363410
Title: Quantifying the Effects of MagnéVie B6® on Stress and Burnout Among Nurses During the COVID-19 Pandemic: A Randomized Double Blind Placebo-Controlled Trial
Brief Title: Micronutrient Supplement for Nurse Burnout
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nutraceuticals Research Institute (Other)
Collaborators: Opella Healthcare Group SAS, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-04-180
Record Dates: First submitted 2022-04-29; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Burnout, Professional; Stress, Psychological
MeSH Terms: conditions — Burnout, Professional; Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MagnéVie B6® (Experimental): Each film coated tablet contains 100mg magnesium citrate and 10mg pyridoxine hydrochloride.
  Interventions: Dietary Supplement: MagnéVie B6®
- Placebo (Placebo Comparator): Each identical film coated tablet contains inert materials.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MagnéVie B6® — micronutrient supplement
  Arms: MagnéVie B6®
Other: Placebo — placebo supplement
  Arms: Placebo

SUMMARY:
The purpose of this study is to confirm and quantify the ability of an 8-week intervention with a supplement containing magnesium citrate and vitamin B6 to reduce anxiety, stress, and burnout among nurses working full time in hospitals and urgent care centers during the COVID-19 Pandemic.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants woh meet the eligibility criteria will provide written informed consent. They will then be randomized in a 1:1 ratio to either MagnéVie B6® or a placebo group. The assigned product will be consumed 3 times daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Woman aged 20-59
* Lives in the United States
* In good general health as evidenced by medical history
* Stress subscale score from the DASS > =22
* Ability to take oral medication and be willing to commit to taking 3 tablets a day for 8 weeks.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of MagnéVie B6® administration
* Employed full time as a nurse in a hospital, primary, or urgent care center that treats COVID-19 patients. Full time is defined as 35 hours or more each week.
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

* Current use of the following pharmaceuticals: bisphosphonates, calcium channel blockers, digoxin, aminoglycoside antibiotics, ketamine, levodopa/carbidopa, gabapentin, potassium sparing diuretics, quinolone antibiotics, skeletal muscle relaxants, sulfonylureas, tetracycline antibiotics, amiodarone, antihypertensives, or antiepileptic drugs (including phenytoin, valproic acid, carbamazepine, phenobarbital).
* Pregnancy, trying to conceive or breastfeeding
* Known allergic reactions to any components of the supplement including magnesium citrate anhydrous, pyridoxine hydrochloride, lactose anhydrous, magnesium stearate, hypromellose, macrogol 6000 titanium dioxide, or talc
* Positive COVID-19 test within 60 days of the study period
* COVID vaccine of any type scheduled during the intervention period or the week prior to the start of the study
* Current diagnosis or lifetime history of a bleeding disorder, kidney disease, or neuromuscular disease
* Recent dramatic weight changes (10% change in body weight in the last 6 months)
* Existing usage of a magnesium or vitamin B6 supplement

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self representation of gender identity
Enrollment: 88 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Scores on the Depression Anxiety Stress Scale (DASS-42), stress sub-score after 8 weeks of intervention as compared to a control group, after controlling for baseline scores. | 8 weeks
  The Depression Anxiety Stress Scale (DASS) 42 is a validated self report measure assessing depression, stress, and anxiety. The scale includes 42 total questions with 14 in each subscale. Higher scores indicate higher severity.

SECONDARY OUTCOMES:
Scores on the State-Trait Anxiety Inventory after 8 weeks of intervention as compared to a control group, after controlling for baseline scores. | 8 weeks
  The STAI is a validated, self reporting instrument assessing anxiety. Possible scores range from 20-80 with higher scores indicating lower quality wellbeing. The instrument contains 40 items.
Scores on the Maslach Burnout Inventory for Health Personnel after 8 weeks of intervention as compared to a control group, after controlling for baseline scores. | 8 weeks
  The Maslach Burnout Inventory for Health Personnel measures the impact of stress specifically among healthcare professionals. It includes emotional exhaustion, loss of feeling towards patients, and the loss of feelings of competence and accomplishment in work. Items are scored on a 1-7 scale and combined by domain, with higher scores indicating greater levels of burnout.
Number of participants with adverse events. | 8 weeks
  All AEs will be documented during the study, as they occur.

OTHER OUTCOMES:
Scores on the DASS-42 total, anxiety, and depression sub-scores after 8 weeks of intervention as compared to a control group, after controlling for baseline scores. | 8 weeks
  The Depression Anxiety Stress Scale (DASS) 42 is a validated self report measure assessing depression, stress, and anxiety. The scale includes 42 total questions with 14 in each subscale. Higher scores indicate higher severity.
Scores on the Magnesium Deficiency Questionnaire (MDQ-62) after 8 weeks of intervention as compared to a control group, after controlling for baseline scores. | 8 weeks
  The MDQ-62 contains 62 self report items which assess magnesium deficiency symptoms in the body. Higher scores indicate a greater probability of magnesium deficiency.
Scores on the DASS-42, MBI-HSS, and STAI after 4 weeks of intervention as compared to a control group, after controlling for baseline scores. | 4 weeks
  The Depression Anxiety Stress Scale (DASS) 42 is a validated self report measure assessing depression, stress, and anxiety. The scale includes 42 total questions with 14 in each subscale. Higher scores indicate higher severity.
Cortisol awakening response after 8 weeks of intervention as compared to a control group after controlling for baseline scores. | 8 weeks
  Salivary cortisol samples will be collected to measure the awakening response. This includes cortisol samples immediately after waking, followed by 30 minutes after waking, for 2 consecutive days. This will be done at baseline and posttest.

CONTACTS AND LOCATIONS:
Overall Officials: JESSIE HAWKINS, PhD, Principal Investigator — Nutraceuticals Research Institute
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No